CLINICAL TRIAL: NCT02092168
Title: Single-dose and Steady-state Pharmacokinetics of BIA 9-1067 and Its Metabolites in Healthy Male Elderly Subjects Compared With Those in Healthy Male Young Subjects
Brief Title: Pharmacokinetics of BIA 9-1067 and Its Metabolites in Healthy Male Elderly Subjects and in Healthy Male Young Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-105
Record Dates: First submitted 2012-01-20; First posted 2014-03-20 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson Disease
Keywords: Opicapone; BIAL
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIA 9-1067 30 mg (once daily) - Elderly Subjects (Experimental): BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 30 mg (once daily) - Young Subjects (Experimental): BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  Interventions: Drug: BIA 9-1067

INTERVENTIONS:
Drug: BIA 9-1067
  Other Names: Opicapone, OPC

SUMMARY:
The purpose of this study is to determine the effects of age on the pharmacokinetic (PK) profile of BIA 9-1067 and its metabolites.

DETAILED DESCRIPTION:
Methodology:

Single-centre, open-label, parallel group, non-randomised multiple-dose 7-day study in 12 healthy elderly and 12 healthy younger male subjects.

Duration of treatment:

Each subject participated in the study for approximately 6 weeks. Participation included a screening evaluation within 28 days before inpatient period, a 12 day inpatient period and an end of study visit (ESV) 7 to 10 days after the discharge from the Unit.

The study design followed the recommendations of the CPMP/ICH/379/95 (ICH Topic E7) Note for Guidance on Studies in Support of Special Populations: Geriatrics, namely in the inclusion of subjects aged 65 years or older and contemplating single-dose and steady-state PK profiles. As the primary endpoint of the study was to characterize the pharmacokinetic profile of BIA 9-1067 and its metabolites in different parallel groups, there was no need to implement blinding procedures or to include a control group. Consequently, the trial was an open label study. Healthy subjects rather than patients with Parkinson's disease have been chosen as the study population, due to the lack of over-toxicity of the drug and an acceptable risk-benefit ratio. This allowed for a better interpretation of the study results, as there were no confounding factors resulting from changes in disease state and or concomitant medications.

The subjects were given a screening number after signing the informed consent by chronological order of inclusion in each group (young/elderly).

ELIGIBILITY:
Inclusion Criteria:

All subjects (young and elderly):

1. A signed and dated informed consent form before any study-specific screening procedure is performed.
2. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead electrocardiogram (ECG).
3. Non-smoker or smoker of fewer than 10 cigarettes per day as determined by history. Had to be able to abstain from smoking during the inpatient stay.
4. With a body mass index (BMI) between 19 and 30 kg/m2, inclusive.

   Young subjects only:
5. Males aged between 18 and 40 years, inclusive.

   Elderly subjects only:
6. Males older than 65 years, inclusive.

Exclusion Criteria:

All subjects (young and elderly):

General

1. Subjects who had participated in a clinical trial with an investigational drug within the 90 days prior to screening.
2. Subjects who were likely to be noncompliant with the protocol, or who were felt to be unsuitable by the Investigator for any other reason.
3. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
4. Positive findings of urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-ethylenedioxymethamphetamine; ecstasy]).

   Medical History
5. Any significant cardiovascular, hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes,), immunological, dermatological, haematological, neurological, or psychiatric disease and history thereof.
6. Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study Day 1.
7. History of drug abuse within 1 year before study Day 1.
8. History of alcoholism within 1 year before Day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g).
9. History of any clinically important drug allergy.
10. Had previously received BIA 9-1067.

    Prohibited treatments and dietary restrictions
11. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 hours before study Day 1.
12. Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before IMP administration.
13. Donation of blood (i.e. 450 ml) within 60 days before study Day 1.

    Young subjects only:

    Prohibited treatments and dietary restrictions
14. Prohibited Treatments: use of any investigational drug within 90 days (young and elderly subjects) or prescription drug within 30 days before investigational medical product (IMP) administration.

    Elderly subjects only:

    Prohibited treatments and dietary restrictions
15. For elderly subjects, previously prescribed medications that do not interfere with absorption, distribution, metabolism, and excretion or safety/tolerability evaluation of BIA 9-1067 and adrenal or renal function were allowed if the dose regimen had been stable for at least 4 weeks and was expected to remain stable throughout the study. Such concomitant medications was reviewed and mutually agreed upon by the sponsor and the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrício SOARES-DA-SILVA, MD, PhD, Study Director — BIAL - Portela & Ca S.A.
Locations (1):
- BIOTRIAL, Rueil, Malmaison, France

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067 30 mg (QD) - Elderly Subjects: BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  BIA 9-1067 30 mg (QD) - Elderly Subjects
- BIA 9-1067 30 mg (QD) - Young Subjects: BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  BIA 9-1067 30 mg (QD) - Young Subjects
Period: Overall Study
Arm/Group | BIA 9-1067 30 mg (QD) - Elderly Subjects | BIA 9-1067 30 mg (QD) - Young Subjects
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BIA 9-1067 30 mg (Once Daily) - Elderly Subjects: BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  BIA 9-1067 30 mg (once daily) - Elderly Subjects
- BIA 9-1067 30 mg (Once Daily) - Young Subjects: BIA 9-1067 was administered as oral doses of 30 mg (5 and 25 mg capsules), once-daily in the morning, during 7 days.
  BIA 9-1067 30 mg (once daily) - Young Subjects
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects | BIA 9-1067 30 mg (Once Daily) - Young Subjects | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 12 | 12
  >=65 years | 12 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration
Description: Cmax (BIA 9-1067) - maximum plasma concentration of BIA 9-1067
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects | BIA 9-1067 30 mg (Once Daily) - Young Subjects
Number analyzed (Participants) | 12 | 12
ng/mL
  Day 1 | 407.4 (81.1) | 391.1 (138.0)
  Day 7 | 439.6 (127.5) | 382.0 (146.6)

2. Primary Outcome: Tmax - Time to Reach Cmax
Description: Tmax - Time to reach maximum plasma concentration of BIA 9-1067
Time Frame: Day 1 and Day 7
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects | BIA 9-1067 30 mg (Once Daily) - Young Subjects
Number analyzed (Participants) | 12 | 12
hours
  Day 1 | 2.0 [1.0 to 4.0] | 2.2 [0.5 to 3.0]
  Day 7 | 2.3 [0.5 to 4.0] | 2.7 [1.5 to 4.0]

3. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration
Description: AUC0-t - Area under the plasma concentration-time curve of BIA 9-1067 from time 0 to last observed concentration
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects | BIA 9-1067 30 mg (Once Daily) - Young Subjects
Number analyzed (Participants) | 12 | 12
ng.h/mL
  Day 1 | 1265.9 (240.6) | 1204.1 (474.7)
  Day 7 | 1413.65 (451.3) | 1112.3 (338.4)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects | BIA 9-1067 30 mg (Once Daily) - Young Subjects
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 30 mg (Once Daily) - Elderly Subjects (N=12) | BIA 9-1067 30 mg (Once Daily) - Young Subjects (N=12)
Influenza like illness (General disorders) | 0 | 1
Bronchitis lymphangitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other